CLINICAL TRIAL: NCT01171508
Title: Circadian Disturbances After Breast Cancer Surgery
Acronym: CIRCA
Status: Completed | Type: Observational
Sponsor: Melissa Voigt Hansen (Other)
Responsible Party: Sponsor-Investigator, Melissa Voigt Hansen, M.D. ph.D student, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: MVH-02
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Circadian Rhythm Disorders; Anxiety; Breast Cancer
Keywords: Circadian Rhythm Disorders; Breast Neoplasms Surgery; Sleep; Heart Rate
MeSH Terms: conditions — Chronobiology Disorders; Anxiety Disorders; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients: 12 breast cancer patients aged 30-70 years undergoing a lumpectomy at Herlev Hospital. ASA score I-III.
  Interventions: Device: Wrist-Actigraph - Octagonal Basic Motionlogger, Ambulatory monitoring Inc, New York, USA; Device: Polysomnograph - Embla A10 (Medcare, Reykjavik, Iceland); Device: Holter monitor - Medilog AR12 (Oxford Instruments, Oxford, England); Procedure: Urine 6-sulphatoxymelatonin (aMT6s); Other: Karolinska Sleepiness Scale; Other: Visual Analog Scale and 10 point-scales to measure fatigue, general well-being, subjective sleep and pain; Other: Sleep-diary

INTERVENTIONS:
Device: Wrist-Actigraph - Octagonal Basic Motionlogger, Ambulatory monitoring Inc, New York, USA — Wrist-Actigraph to be worn on the non-dominant arm on day 0-3-17 of the study.
Device: Polysomnograph - Embla A10 (Medcare, Reykjavik, Iceland) — Polysomnography on day 0-3-17 of the study. This is a portable polysomnograph with 16 digital channels for recording of electroencephalogram (EEG), electrooculograph (EOG) and electromyograph (EMG).
Device: Holter monitor - Medilog AR12 (Oxford Instruments, Oxford, England) — Holter monitoring on day 0-3-17 of the study. Measurements are done by superficial skin-electrodes placed after standardised rules from the producer of the device.
Procedure: Urine 6-sulphatoxymelatonin (aMT6s) — Urine sampling for measurement of the primary metabolite of melatonin - 6-sulphatoxymelatonin (aMT6s) will be done on day 0-3-17 of the study. The analysis will be done by a radioimmunoassay.
Other: Karolinska Sleepiness Scale — Karolinska Sleepiness Scale to measure sleepiness will be filled out twice a day every day of the entire study period of 17 days.
Other: Visual Analog Scale and 10 point-scales to measure fatigue, general well-being, subjective sleep and pain — Visual Analog Scale and 10 point-scales to measure fatigue, general well-being, subjective sleep and pain will be filled out twice a day everyday of the study period of 17 days.
Other: Sleep-diary — Sleep-diary to measure subjective sleep quantity will be completed every morning and after every nap in the day.

SUMMARY:
The purpose of this study is to investigate circadian disturbances after breast cancer surgery by means of monitoring sleep and heart-rate variability, by measuring a metabolite of melatonin in urine and by questionnaires and a sleep-diary.

DETAILED DESCRIPTION:
An increasing number of studies have shown that circadian variation in the excretion of hormones, the sleep-wake cycle, the core body temperature, the tone of the autonomic nervous system and the activity rhythm are important both in health and disease processes. More attention is being paid towards the circadian variation in endogenous rhythms in relation to surgery and whether this can affect postoperative recovery, morbidity and mortality.

Studies have been done on circadian disturbances after major and minor surgery but never in relation to breast cancer surgery.

This study will investigate circadian disturbances in this specific group of patients by using Actigraphy, Polysomnography (PSG), Holter-monitoring (HRV), the primary metabolite of melatonin in urine 6-sulfatoxymelatonin (aMT6s), questionnaires and a sleep-diary.

ELIGIBILITY:
Inclusion Criteria:

* women, age 30-70, with breast cancer who are admitted for a lumpectomy at Herlev Hospital
* ASA score I-III

Exclusion Criteria:

* Known sleep apnea
* Pre-operative treatment with beta-blockers
* Diabetes Mellitus
* Known pre-operative depressive illness or dementia
* Previous or current cancer
* Known medically treated sleep-disorder (insomnia, restless legs etc)
* Shift-work
* Daily alcohol intake of more than 5 units
* Pre-operative treatment with psychopharmacological drugs, opioids or anxiolytics (including all sleeping pills)
* Predicted bad compliance
* Pregnant or breast-feeding
* Pre- or post-operative complications or events which are expected to increase morbidity or pain the first post-operative days.
* Missing written consent
* Pre-operative MMSE score less than 24
* Urine or fecal incontinence

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Breast Surgery at Herlev University Hospital in Copenhagen
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Preoperative sleep architecture of breast cancer patients | 1 day preoperatively
  Sleep architecture measured by Polysomnography (awake, stadium I-IV, REM sleep, sleep latency, awakenings).
Postoperative sleep architecture of breast cancer patients (early phase) | The first postoperative night
  Sleep architecture measured by Polysomnography (awake, stadium I-IV, REM sleep, sleep latency, awakenings)
Postoperative sleep architecture of breast cancer patients (late phase) | The 14th postoperative night
  Sleep architecture measured by Polysomnography (awake, stadium I-IV, REM sleep, sleep latency, awakenings)
Sleep quality, fatigue, well-being and pain. | 1 day preoperatively till 14 days postoperatively
  Fatigue, generel well-being, subjective sleep and pain scores on a Visual Analog Scale - questionnaires filled out daily. Sleepiness measured by Karolinska Sleepiness Scale. A sleep-diary recording sleep quantity of day and night sleep.
Preoperative melatonin levels and amplitude | 1 day preoperatively
  Excretion of aMT6s in urine. Urine will be collected from 23-07, quantified and 2 samples will be taken to measure aMT6s.
Postoperative melatonin levels and amplitude (early phase) | The first postoperative night
  Excretion of aMT6s in urine. Urine will be collected from 23-07, quantified and 2 samples will be taken to measure aMT6s.
Postoperative melatonin levels and amplitude | The 14th postoperative night
  Excretion of aMT6s in urine. Urine will be collected from 23-07, quantified and 2 samples will be taken to measure aMT6s.
Sleep architecture | 1 day preoperatively till 14 days postoperatively
  Actigraphy (total minutes asleep, sleep effectiveness, sleep latency, awakenings). A wrist actigraph wil be worn from 1 day preoperatively and taken off on the 14th postoperative day.

SECONDARY OUTCOMES:
Preoperative heart-rate variability of breast cancer patients | 1 day preoperatively
  Heart-rate variability measured by Holter monitor and a following analysis of frequency domain parameters.
Postoperative heart-rate variability of breast cancer patients (early phase) | The first postoperative night
  Heart-rate variability measured by Holter monitor and a following analysis of frequency domain parameters.
Postoperative heart-rate variability of breast cancer patients (late phase) | The 14th postoperative night
  Heart-rate variability measured by Holter monitor and a following analysis of frequency domain parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa V Hansen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Copenhagen, Denmark